CLINICAL TRIAL: NCT01052818
Title: Therapeutic and Prognostic Impact of Circulating Tumor Cells in Peripheral Blood in Patients With Non Small-cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Oscar Arrieta Rodriguez, CONACyT
Other Study IDs: INCAN/OfCA204/SO151/CB451/09; 87453 (Other: National Counsil of Science and Technology)
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Circulating Tumor Cells
Keywords: Non small-cell lung cancer; Circulating tumor cells; Carcinoembryonic antigen; Cytokeratin
MeSH Terms: conditions — Neoplastic Cells, Circulating; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples are collected were the cell pellet are collected from centrifugation, lysed by TRIzol method to get RNA. The RNA is retrotranscribed to cDNA in order to quantify cytokeratin (CK) 19, 18 and carcinoembrionic antigen which are markers of epithelial cells presumambly coming form the tumor.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stage IV NSCLC: Stage IV non small-cell lung cancer patients will be recruited for this protocol

SUMMARY:
The purpose of the study is to evaluate the association between the number of circulating tumor cells and response to treatment in non small-cell lung cancer patients

DETAILED DESCRIPTION:
In spite of technological advantages in diagnosis and treatment, lung cancer remains one of the most deadly malignant neoplasias. Moreover, there are no markers for monitoring response to treatment. The objective of the study is to associate the number of circulating tumor cells (CTC) before and after treatment and correlate it with tumor response rate, progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic diagnosis of non small-cell lung cancer
* Clinical stage IV
* ECOG functional status 0 or 1
* No renal function alteration (GFR >50%)
* No hepatic function alteration (ALT and AST less than 2 times its normal value)
* Leucocytes more than 2,000/mcl
* Hemoglobin more than 10mg/dL
* Platelets more than 100,000/mcl

Exclusion Criteria:

Non-advanced disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced non small-cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Response rate, progression-free survival and over-all survival | 4 years

SECONDARY OUTCOMES:
Quantification of CTCs | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD, Principal Investigator — National Counsil of Science and Technology
Locations (1):
- National Institute of Cancerologia, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Arrieta O, Pineda B, Muniz-Hernandez S, Flores D, Ordonez G, Borbolla-Escoboza JR, Orta D. Molecular detection and prognostic value of epithelial markers mRNA expression in peripheral blood of advanced non-small cell lung cancer patients. Cancer Biomark. 2014;14(4):215-23. doi: 10.3233/CBM-140394. PMID 24934364